CLINICAL TRIAL: NCT00284232
Title: Randomized Controlled Trial Studying the Metabolic Effects of Accurate Blood Sugar Results and Education in Type 1 Diabetes
Brief Title: Metabolic Effects of Accurate Blood Sugar Results and Education in Type 1 Diabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Helse Stavanger HF (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: Measure 2004
Record Dates: First submitted 2006-01-27; First posted 2006-01-31 (Estimated); Last update posted 2015-07-28 (Estimated); Status verified 2015-07

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: HbA1c; Self-monitoring blood glucose (SMBG); Diabetes treatment; quality of care
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Use and interpretation of blood glucose results
Drug: Insulin dosing based on SMBG chart and education

SUMMARY:
A randomized controlled trial in patients with type 1 diabetes, assessing the metabolic effects of accurate blood sugar results and education. A systematic approach in self-monitoring blood glucose will improve metabolic control in type 1 diabetes patients. Education in SMBG combined with a high analytical quality instrument for SMBG, introduced in a systematic and thorough way will improve HbA1c by 0,5% and keep it over a period of 9 months.

DETAILED DESCRIPTION:
* Written informed consent 130 patients with type 1 diabetes to be included
* age 18-70
* HbA1c of 8% or higher, variation in HbA1c over the last 18 months sholuld be <1,5%
* Treated with multiple insulin injections or insulin pumps
* Variation in weight less than 5kg within last year
* Using SMBG on a daily basis
* Mental capacity and stability to participate
* No hypoglycemia unawareness
* No likelihood that patient will drop out or not perform according to protocol
* Continious recruitment from the outpatient clinic at Stavanger University Hospital from October 2004-October 2005
* 9 months follow-up
* Possible 12 month extension after initial
* Intervention group receives new SMBG instrument, education and advice on treatment changes at baseline, 1,2,3,6 and 9 months. Control group continues regular care following national guidelines of Norway. This includes visits usually every 3-6 months at the outpatient clinic and possibly with their GP in addition.

ELIGIBILITY:
Inclusion Criteria:

* Hba1c 8% or higher, less than 1,5% variation within last year
* Age 18-70
* Multiinjections or insulin pumps
* Stable weight (<5kg variation last year)
* Mentally stable

Exclusion Criteria:

* Hypoglycemia unawareness
* Mental incapacity

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140
Dates: Start 2004-10; Primary Completion 2006-08 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
HbA1c % | 9 months

SECONDARY OUTCOMES:
Hypoclycemic events | 9 months
Measurement quality of blood glucose instrument | 9 months
Frequency of SMBG | 9 months
Satisfaction | 9 months
New learning points for patients | 9 months
Confidence in new instrument quality | 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Svein Skeie, MD PhD, Principal Investigator — Stavanger Health Research
Locations (1):
- Stavanger University Hospital, Stavanger, Norway